CLINICAL TRIAL: NCT01478204
Title: An Observational Epidemiological Study on Evaluation of Sleep Quality in Patients With Mild to Moderate Alzheimer's Disease in Clinical Practice
Brief Title: A Study to Evaluate Sleep Quality in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017509; GALALZ4037 (Other: Janssen-Cilag S.A., Spain)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Sleep quality; Anticholinesterase drugs
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate sleep quality in patients with mild to moderate Alzheimer's disease treated with anticholinesterase drugs in clinical practice.

DETAILED DESCRIPTION:
This is an epidemiological (the study of health-related states or events in specific populations) study of patients with mild to moderate Alzheimer's who have been treated previously with anticholinesterase drugs (class of drugs that act in the central nervous system) up to a maximum of fifteen days. The data for each patient will be recorded on two occasions; first at a baseline visit and then at a follow-up visit at 3 months. At the baseline visit, after the patient or his/her legal representative has given written informed consent, each participating neurologist will use the study questionnaire to collect patient sociodemographic characteristics (characteristics such as age, years of education, race, sex, religion, birthplace, income, occupation, geographic location, among others), medical history and diagnosis of Alzheimer's disease. The neurologist will also record treatment for Alzheimer's disease and concomitant hypnotic medications (simultaneous use of medications that induce sleep) and evaluate the patient using two scales: the Pittsburgh Sleep Quality Index (PSQI) to record sleep disturbances and the Epworth Sleepiness Scale to determine the level of daytime sleepiness. Alzheimer treatment and concomitant hypnotic medications will be recorded again at the follow-up visit. Patient sleep quality using the PSQI and daytime sleepiness using the Epworth scale will also be evaluated again at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent diagnosis of possible or probable Alzheimer's disease (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA criteria) within a maximum of 60 days before the baseline visit.
* Patients with mild or moderate Alzheimer's disease, defined by a Mini-Mental State Exam (MMSE) score between 11 and 25.
* Patients whose caregivers are sufficiently informed of the patients' state and if possible live with the patient.
* Patients who are capable of attending a second clinic visit with their accompanying person 3 months later, based on the clinical practice of the investigator.
* Patients and/or legal representatives who have given and signed written informed consent.

Exclusion Criteria:

* Patients who have psychotic manifestations.
* Patients who have clinically significant sleep disorder (sleep apnea syndrome, restless leg syndrome).
* Patients treated with memantine.
* Patients and/or legal representatives who refuse to give written informed consent to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the neurology clinic of participating centers throughout Spain who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Sleep disturbances measures by Scores on the Pittsburgh Sleep Quality Index (PSQI) Scale | Up to 3 months
  The PSQI consists of 19 self-rated questions which assesses sleep quality and disturbances over 1-month time interval. The 19 questions assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and the frequency and severity of specific sleep-related problems. These 19 items are grouped into seven components scores, each weighted equally on a 0-3 scale. The seven components scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
The Level of Daytime Sleepiness determined by the Scores on the Epworth Sleepiness Scale | Up to 3 months
  The Epworth Sleepiness Scale measures how likely, from 0 (would never take a nap) to 3 (high change of dozing), the patient is to doze off or fall asleep in common everyday situations. The scores for a total of eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A., Spain Clinical Trial, Study Director — Janssen-Cilag, S.A.